CLINICAL TRIAL: NCT06012734
Title: Phase Ib Study With the Combination of LB-100 (PP2A Inhibitor) and Atezolizumab (PD-L1 Inhibitor) in Metastatic Colorectal Cancer Patients - The CoLBAt Trial
Brief Title: LB-100 (PP2A Inhibitor) and Atezolizumab (PD-L1 Inhibitor) in Metastatic Colorectal Cancer Patients
Acronym: CoLBAt
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N22CLB
Record Dates: First submitted 2023-07-21; First posted 2023-08-25 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Microsatellite-stable Colorectal Cancer
Keywords: Gastrointestinal Neoplasms; Colorectal cancer; Metastatic colorectal cancer; Microsatellite stable; Immune checkpoint inhibitors
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms | interventions — LB100; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LB-100 plus atezolizumab (Experimental): LB-100 IV over 15 minutes on day 1 and day 3 Atezolizumab IV over 30-60 minutes on day 1 Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: LB-100; Drug: Atezolizumab

INTERVENTIONS:
Drug: LB-100 — IV on day 1 and day 3
  Other Names: PP2A inhibitor LB-100
Drug: Atezolizumab — IV on day 1
  Other Names: Tecentriq

SUMMARY:
This Phase Ib trial studies the side effects and best dose of LB-100 when given with atezolizumab for the treatment of patients with metastatic microsatellite stable colorectal cancer. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of the tumor to grow and spread. LB-100 has been shown to make anticancer drugs work better at killing cancer. LB-100 blocks a protein on the surface of cells called PP2A. Blocking this protein increases the stress signals for the tumor cells that express PP2A. Giving atezolizumab in combination with LB-100 may work better to treat metastatic colorectal cancer patients as the cancer cells that experience increased stress signals are more susceptible for the immunotherapy.

DETAILED DESCRIPTION:
The goal of this Phase Ib monocenter, open-label, non-randomized clinical trial is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of the combination of LB-100 and atezolizumab in patients with metastatic microsatellite stable colorectal cancer.

This study will consist of a dose escalation phase and a dose expansion phase. The dose escalation phase is designed to find the recommended phase II dose of LB-100 in combination with atezolizumab standard dosage of 1200 mg. The dose expansion phase further explores the clinical activity, safety, tolerability and pharmacokinetics/dynamics of LB-100 combined with atezolizumab.

LB-100 will be administered intravenously on day 1 and day 3 of every 21-day cycle.

Atezolizumab 1200 mg will be administered intravenously on day 1 of every 21-day cycle, which is the labelled dose as monotherapy.

Clinical assessments will be performed routinely to monitor safety. Anti-tumor activity will be measured by CT scan according to RECIST version 1.1 criteria. Tumor biopsies will be obtained for exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF);
2. Age ≥ 18 years at time of signing ICF;
3. Ability to comply with the study protocol;
4. Histological or cytological confirmed colorectal cancer;
5. Immunohistochemically confirmation of microsatellite stable (MSS) phenotype;
6. Disease progression during treatment with standard of care;
7. Measurable disease per Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1). Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation;
8. Able and willing to undergo blood sampling and tumour biopsies at baseline, if no adequate archival material is available, and during therapy;
9. Availability of representative tumor specimen for exploratory biomarker research;
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
11. Life expectancy of at least 3 months;
12. Negative HIV test at screening. Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/µL, and have an undetectable viral load;
13. Negative hepatitis B test at screening;
14. Negative hepatitis C virus test at screening;
15. Adequate hematologic and end-organ function as defined by:

    * Absolute neutrophil (segmented and bands) count ≥1.0×109/L
    * Lymphocyte count ≥0.5×109/L
    * Platelets≥100×109/L
    * Hemoglobin ≥5.6 mmol/L
    * AST≤2.5×ULN
    * ALT≤2.5×ULN
    * AP ≤2.5×ULN
    * Bilirubin ≤1.5×ULN
    * Estimated glomerular filtration rate ≥50 mL/min by CKD-EPI
    * Albumin ≥25 g/L
    * INR ≤1.5×ULN
    * aPTT ≤1.5×ULN
16. Negative pregnancy test (urine or serum) for female patients with childbearing potential.

Exclusion Criteria:

1. Unable to follow study procedures;
2. Patients using prohibited medication;
3. Any unresolved grade ≥ 2 toxicities related to prior treatments (excluding alopecia) according to CTCAE version 5.0;
4. Symptomatic or actively progressing central nervous system (CNS) metastases. Asymptomatic patients with treated or untreated CNS lesions are eligible, provided that all of the following criteria are met:

   * Measurable disease, per RECIST v1.1, must be present outside the CNS;
   * The patient has no history of intracranial haemorrhage or spinal cord haemorrhage;
   * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment;
   * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease;
   * If the patient is receiving anti-convulsant therapy, the dose is considered stable;
5. History of leptomeningeal disease;
6. Uncontrolled tumor-related pain. Patients requiring pain medication must be on a sta-ble regimen at study entry;
7. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures. Patients with indwelling catheters are allowed;
8. Uncontrolled symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium >12 mg/dL, or corrected calcium greater than ULN);
9. Active or history of auto-immune disease or immune deficiency;
10. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field is permitted;
11. Active tuberculosis;
12. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina;
13. Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study;
14. History of malignancy within 2 years prior to initiation of study treatment, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%);
15. Severe infection within 4 weeks prior to initiation of study treatment;
16. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics are eligible for the study;
17. Prior allogeneic stem cell or solid organ transplantation;
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications;
19. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab;
20. Current treatment with anti-viral therapy for HBV;
21. Treatment with investigational therapy within 28 days prior to initiation of study treat-ment;
22. Prior treatment with CD137 agonists or immune checkpoint blockade therapies;
23. Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives prior to initiation of study treatment;
24. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment;
25. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins;
26. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the Atezolizumab formulation;
27. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The RP2D of LB-100 when given in combination with standard doses of atezolizumab | up to 2 years

SECONDARY OUTCOMES:
Disease control rate | 6 months
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Objective response rate | 6 months
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of overall response | up to 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Progression free survival | up to 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Overall survival | Assessed up to 2 years
  The time from the first dose of study treatment to the time of death from any cause. Patients who are still alive at the time of analysis will be censored at the time of their last study assessment (for active patients) or at the last date know alive (for patients in follow-up).
Observed plasma concentrations of LB-100, its active metabolite endothall and atezolizumab | Prior to initial dose, on day 1, day 2, day 3, day 8, day 15 and prior to second cycle. Each cycle is 21 days
  Blood samples are obtained and plasma concentrations of LB-100, endothall and atezolizumab are measured
Area under the plasma-time concentration curve of LB-100, its active metabolite endothall and atezolizumab | Prior to initial dose, on day 1, day 2, day 3, day 8, day 15 and prior to second cycle. Each cycle is 21 days
  Blood samples are obtained and plasma concentrations of LB-100, endothall and atezolizumab are measured
Elimination half-life of LB-100, its active metabolite endothall and atezolizumab | Prior to initial dose, on day 1, day 2, day 3, day 8, day 15 and prior to second cycle. Each cycle is 21 days
  Blood samples are obtained and plasma concentrations of LB-100, endothall and atezolizumab are measured
Total body clearance of LB-100, its active metabolite endothall and atezolizumab | Prior to initial dose, on day 1, day 2, day 3, day 8, day 15 and prior to second cycle. Each cycle is 21 days
  Blood samples are obtained and plasma concentrations of LB-100, endothall and atezolizumab are measured
The incidence and severity of adverse events | Up to 2 years
  As assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
The incidence of dose-limiting toxicity | 21 days
  As assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

OTHER OUTCOMES:
Serine/threonine hyperphosphorylation in peripheral white blood cells | Blood sample cycle 1 day 1. Each cycle is 21 days.
  Western Blots to evaluate serine/threonine hyperphosphorylation in peripheral white blood cells
Mismatch repair deficiency status | Before start of treatment and one on treatment biopsy at Cycle 3 day 3. Each cycle is 21 days
  Immunohistochemistry for mismatch repair proteins
Concentration of LB-100 and endothall in tumor tissue | On treatment biopsy at Cycle 3 day 3. Each cycle is 21 days
  To evaluate pharmacodynamic biomarkers of LB-100

CONTACTS AND LOCATIONS:
Overall Officials: Neeltje Steeghs, MD, PhD, Principal Investigator — The Netherlands Cancer Institute - Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No